CLINICAL TRIAL: NCT05350319
Title: Prospective Comparison of Simulated Low Dose Computed Tomography to Conventional Dose Computed Tomography for the Evaluation of Glenoid Anatomy in Shoulder Arthroplasty
Brief Title: Prospective Low Dose CT for Total Shoulder Arthroplasty/Reverse Shoulder Arthroplasty
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00108187
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Shoulder Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients planning for total or reverse shoulder arthroplasty: Adult patients who are planning to undergo a total or reverse shoulder arthroplasty
  Interventions: Radiation: A low-dose CT scan of the shoulder
- Retrospective group of patients who have already undergone preoperative planning: Retrospective cohort of patients who have undergone preoperative planning with a conventional shoulder CT for total or reverse shoulder arthroplasty.

INTERVENTIONS:
Radiation: A low-dose CT scan of the shoulder — Briefly, a conventional CT scan will be conducted, with scan images representing a reconstruction of simultaneous scans at two sensors. L-CT images will be derived from single source data (ie the scan data gathered by one of the emitters rather than a reconstruction from both).
  Groups: Patients planning for total or reverse shoulder arthroplasty

SUMMARY:
This study is a prospective, departmental funded study examining the outcomes of simulated Low Dose CT scans compared to Conventional Dose CT scans in patients who present to Duke University for total shoulder arthroplasty or reverse shoulder arthroplasty.

DETAILED DESCRIPTION:
The purpose of this study is to compare the use of a conventional dose computed tomography scan (C-CT) to a simulated low dose computed tomography scan (L-CT) for preoperative planning in patients who are anticipated to undergo a total shoulder arthroplasty (TSA) or reverse shoulder arthroplasty (RSA) with the goal to reduce the radiation exposure to future patients undergoing preoperative planning. L-CT scans for analysis will be obtained prospectively as derived data from a C-CT scan performed on a dual source CT scanner. Briefly, a C-CT scan will be conducted, with scan images representing a reconstruction of simultaneous scans at two sensors. L-CT images will be derived from single source data (ie the scan data gathered by one of the emitters rather than a reconstruction from both). For additional validation, prospectively collected scans will be compared to retrospectively gathered scans of patients of similar demographics (age, sex, BMI) and degenerative changes who underwent a C-CT scan for an anticipated shoulder arthroplasty in the past. The reviewers will investigate the following outcome measures including 1) Are L-CT images of sufficient quality to be used for preoperative planning 2) Can accurate measurements including glenoid inclination, version, implant selection and humeral head subluxation be made on L-CT images 3) Do proposed treatment plans change with the use of L-CT relative to the chosen plans base on C-CT images. The investigators hypothesize L-CT images will be of sufficient image quality for diagnostic purposes, with similar measurements, and treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are planned to undergo total or reverse shoulder arthroplasty
* Subject must be 18 years or older
* Subjects who have capacity to give informed consent

Exclusion Criteria:

* Subjects who are pregnant
* Subjects under the age of 18
* Subjects who do not have the capacity to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All individuals who are scheduled for a shoulder CT for the purpose of preoperative planning for a total shoulder arthroplasty are eligible to be included in this study assuming they meet the eligibility requirements as listed above.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Low Dose CT Images of Sufficient Pre-operative Planning Quality | Day 1
  Low Dose CT Images will be compared to a standard dose to assess image quality.
Glenoid Version | Day 1
  Representative CT images will be used to measure the version of each shoulder for preoperative purposes.
Glenoid Inclination | Day 1
  Representative CT images will be used to measure the inclination of each shoulder for preoperative purposes.
Humeral Head Subluxation | Day 1
  Representative CT images will be used to measure the humeral head subluxation of each shoulder for preoperative purposes.
Implant Selection | Day 1
  Representative CT images will be used to determine the implant selection for preoperative purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Klifto, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data is not planned to be shared outside of the collaborators of this project within the Duke University Medical Center. The data will only be reviewed by the study personnel listed on the Institutional Review Board (IRB), and not intended to be shared with an external institution or industry.
  However, when submitting data for manuscripts and publication purposes, all data will be deidentified of any public health information. All Protected Health Information (PHI) will be kept in a locked cabinet in the PI's office at Duke University and/or in a protected/encrypted folder in a file separate from the study information. Data will be analyzed by study team members using a computer that is password protected, and stored securely in encrypted Duke servers.
  Study files will be backed up onto Dr. Klifto's folder in a secure server provided to faculty in the Department of Orthopaedic Surgery. The subjects will not be identified in any reports or publications from this study.

REFERENCES:
- [Background] Biswas D, Bible JE, Bohan M, Simpson AK, Whang PG, Grauer JN. Radiation exposure from musculoskeletal computerized tomographic scans. J Bone Joint Surg Am. 2009 Aug;91(8):1882-9. doi: 10.2106/JBJS.H.01199. PMID 19651945
- [Background] Iannotti JP, Weiner S, Rodriguez E, Subhas N, Patterson TE, Jun BJ, Ricchetti ET. Three-dimensional imaging and templating improve glenoid implant positioning. J Bone Joint Surg Am. 2015 Apr 15;97(8):651-8. doi: 10.2106/JBJS.N.00493. PMID 25878309
- [Background] Yu L, Shiung M, Jondal D, McCollough CH. Development and validation of a practical lower-dose-simulation tool for optimizing computed tomography scan protocols. J Comput Assist Tomogr. 2012 Jul-Aug;36(4):477-87. doi: 10.1097/RCT.0b013e318258e891. PMID 22805680
- [Background] Boileau P, Cheval D, Gauci MO, Holzer N, Chaoui J, Walch G. Automated Three-Dimensional Measurement of Glenoid Version and Inclination in Arthritic Shoulders. J Bone Joint Surg Am. 2018 Jan 3;100(1):57-65. doi: 10.2106/JBJS.16.01122. PMID 29298261
- [Background] Tipnis SV, Spampinato MV, Hungerford J, Huda W. Thyroid Doses and Risks to Adult Patients Undergoing Neck CT Examinations. AJR Am J Roentgenol. 2015 May;204(5):1064-8. doi: 10.2214/AJR.14.13102. PMID 25905942
- [Background] Maurer A, Fucentese SF, Pfirrmann CW, Wirth SH, Djahangiri A, Jost B, Gerber C. Assessment of glenoid inclination on routine clinical radiographs and computed tomography examinations of the shoulder. J Shoulder Elbow Surg. 2012 Aug;21(8):1096-103. doi: 10.1016/j.jse.2011.07.010. Epub 2011 Oct 29. PMID 22036540